CLINICAL TRIAL: NCT00906763
Title: Effects of Chocolate on Motor Symptoms of Parkinson's Disease - A Monocenter, Prospective, Observer-blinded Interventional Trial
Brief Title: Effects of Chocolate on Motor Symptoms of Parkinson's Disease
Acronym: ChocoPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Martin Wolz, MD, Dresden University of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EK284112008
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Neurodegenerative Disorders; Biogenic amines; Chocolate; Cocoa
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases | interventions — Chocolate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dark Chocolate (85% cocoa) (Active Comparator): Oral Intake of dark chocolate (85% cocoa) over 15 minutes.
  Interventions: Dietary Supplement: Chocolate
- White chocolate (0% cocoa) (Active Comparator): Oral intake of 200 grams of white chocolate (0% cocoa) over 15 Minutes.
  Interventions: Dietary Supplement: Chocolate

INTERVENTIONS:
Dietary Supplement: Chocolate — A single oral application of 200 grams of chocolate (85% cocoa for arm #1; 0% cocoa for arm #2).

SUMMARY:
Chocolate consumption has long been associated with enjoyment and pleasure. Popular claims confer on chocolate the properties of being a stimulant, relaxant, euphoriant and antidepressant. These possible pharmacological actions might be related to various biogenic amines, such as serotonin, dopamine, tyramine, histamine, phenylethylamine and cannabinoid-like substances. Most amines are metabolized by monoamineoxidase-A (MAO-A) and are therefore unable to pass the blood-brain-barrier. In contrast, phenylethylamine is a direct dopamine releasing ingredient and as a substrate of MAO-B and due to its lipophilic structure even capable to pass the blood-brain-barrier. Within this line, own clinical observations suggested an increased chocolate consumption in patients with Parkinson's disease (PD) compared to healthy subjects and to their pre-disease state.

In a previous study, we assessed the consumption of chocolate and non-chocolate sweets in PD patients and their partners (as household controls) using a self-questionnaire. Consumption of chocolate was significantly higher in PD patients compared to controls, while consumption of non-chocolate sweets was similar in both groups. Our study suggests that chocolate consumption is increased in PD independent of concomitant depressive symptoms measured by BDI-1. Although reasons for increased chocolate consumption in PD remain elusive, it may hypothetically be a consequence of the high content of various biogenic amines as a content of cocoa influencing dopamine metabolism.

Therefore, in the present study we aim to study the effects of dark chocolate with high cocoa content (85%) compared to chocolate without any cocoa (white chocolate) on motor symptoms in PD patients as measured with UPDRS part III (motor score). The principle design of the intervention is similar to the standard pharmacological challenge test for studying effects on motor symptoms in PD (e.g. levodopa challenge test).

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 Years or older
* Idiopathic Parkinson's disease, according to UKBB criteria
* Hoehn & Yahr Score II-III
* 16 Points or more in UPDRS part III scale
* Sufficient ability to follow the study procedure for at least 3 hours
* Ability to give informed consent
* Stable antiparkinsonian medication for at least 4 weeks prior to study inclusion

Exclusion Criteria:

* Psychiatric conditions, severe enough to interfere with study procedures
* motor or affective fluctuations or dyskinesias
* treatment with COMT and/or MAO inhibitors
* Diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-08 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
UPDRS part III | 1 h after intake of study intervention

SECONDARY OUTCOMES:
Biogenic amines in blood | 1 to 3 h after study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wolz, MD, Principal Investigator — Technische Universität Dresden
Locations (1):
- Dresden University of Technology, Medical Faculty, Dresden, Germany

REFERENCES:
- [Background] Wolz M, Kaminsky A, Lohle M, Koch R, Storch A, Reichmann H. Chocolate consumption is increased in Parkinson's disease. Results from a self-questionnaire study. J Neurol. 2009 Mar;256(3):488-92. doi: 10.1007/s00415-009-0118-9. Epub 2009 Mar 13. PMID 19277767